CLINICAL TRIAL: NCT00423618
Title: Randomised Trial of Post-Operative Radiotherapy Given to Adult Patients With Extremity Soft Tissue Sarcoma [VORTEX]
Brief Title: Randomised Trial of Volume of Post-operative Radiotherapy Given to Adult Patients With eXtremity Soft Tissue Sarcoma
Acronym: VORTEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH14490 CRUK-VORTEX; CDR0000526239 (Registry Identifier: PDQ (Physician Data Query)); EU-20678 (Other: NK); ISRCTN76456502 (Registry Identifier: ISRCTN); CRCTU-SA3002 (Other: CR UK Clinical Trials Unit, University of Birmingham)
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; adult synovial sarcoma; adult angiosarcoma; adult epithelioid sarcoma; adult extraskeletal chondrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult fibrosarcoma; adult neurofibrosarcoma; adult alveolar soft-part sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial; Hemangiosarcoma; Chondrosarcoma, Extraskeletal Myxoid; Leiomyosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Fibrosarcoma; Neurofibrosarcoma; Sarcoma, Alveolar Soft Part | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (Active Comparator): Radiotherapy Conventional treatment arm A total of 33 fractions each of 2Gy should be given once a day for 5 days per week over 6 weeks and 3 days in week 7, totalling 66Gy. The first 50 Gy in 25 fractions will be given to CTV1 and subsequent 16 Gy in 8 fractions will be delivered to CTV2.
  Interventions: Radiation: radiotherapy
- Research arm (Experimental): Radiotherapy Research arm A total of 33 fractions each of 2Gy should be given once a day for 5 days per week over 6 weeks and 3 days in week 7, totalling 66Gy. The 66Gy in 33 fractions will be delivered to CTV2 alone. No attempt will be made to include drain/biopsy sites or the surgical scar.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy as adjuvant treatment for adults with soft tissue sarcoma extremities

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving radiation therapy to a smaller area of tissue surrounding the tumor is as effective as giving radiation therapy to a wider area of tissue surrounding the tumor in treating soft tissue sarcoma.

PURPOSE: This randomized phase III trial is studying giving external-beam radiation therapy to a small area of tissue surrounding the tumor to see how well it works compared with giving external-beam radiation therapy to a wider area of tissue surrounding the tumor in treating patients who have undergone surgery for soft tissue sarcoma of the arms, hands, legs, or feet.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if reduced volume adjuvant radiotherapy increases limb function without compromising local control in patients with previously resected extremity soft tissue sarcoma.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the overall level of disability in patients treated with this regimen.
* Determine the disease-free survival and overall survival of these patients.

OUTLINE: This is a randomized, controlled, prospective, multicenter study. Patients are stratified according to tumor grade (1 vs 2 vs 3), adequacy of surgical clearance (R0 vs R1), and treatment center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients undergo external beam radiotherapy (EBRT), including full margins, once daily 5 days a week for 6½ weeks .
* Arm II: Patients undergo EBRT as in arm I but only reduced margins are included.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma meeting the following criteria:

  * Lesion originates in extremity

    * Upper extremity lesions may occur from the medial border of the scapula to tumors as far distal as the finger tips

      * No lesions of the chest wall arising adjacent to the scapula but not originating in the shoulder bone
    * Lower extremity regions include hip girdle tumors commencing at the iliac crest, excluding lesions arising from within the pelvis, and extends to include lesions as far distal as the toes
  * Imaging and pathology from first surgery are required
* Has undergone surgical resection of the tumor within the past 12 weeks

  * No macroscopic tumor in situ after surgery
  * Microscopically irradical surgical margin allowed
  * Excisional biopsy with positive margins or other inadequate surgery (macroscopically involved margins) allowed only after further definitive re-excision
  * Positive margins and no further surgery possible except amputation or major functional loss allowed provided no macroscopic residual disease is present
  * Local recurrence within 3 months of prior surgery (or other treatment) allowed provided patient undergoes subsequent re-excision
* No diagnosis of any of the following:

  * Rhabdomyosarcoma (alveolar or embryonal)
  * Primitive neuroectodermal tumor
  * Soft tissue Ewing's sarcoma
  * Extraskeletal osteosarcoma
  * Aggressive fibromatosis (desmoid tumors)
  * Dermatofibrosarcoma protuberans
  * Gorlin's syndrome
* No regional nodal disease or unequivocal distant metastasis

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No other major medical illness that would preclude study treatment
* No other malignancy except adequately treated nonmelanomatous carcinoma of the skin or in situ carcinoma of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to the local site
* No prior neoadjuvant or adjuvant chemotherapy

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Limb functionality as measured by the Toronto Extremity Salvage Score (TESS) | 2 years
Time to local recurrence | time from randomisation into the trial to the occasion when a local recurrence is confirmed by biopsy. For those patients who are not observed to have a local recurrence during the course of the study, the time to local recu

SECONDARY OUTCOMES:
Soft tissue and bone toxicity as measured by RTOG | 2 years
Disease-free survival | defined in whole days as time from randomisation into the trial to either local or distant recurrence or death (whichever occurs first).
Overall survival | defined in whole days as time from randomisation into the trial to death.
Overall level of disability as measured by the TESS questionnaire | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Robinson, MD, Study Chair — Cancer Research Centre at Weston Park Hospital
Locations (6):
- United Kingdom (6):
  - Royal Orthopedic Hospital NHS Trust, Birmingham, England
  - Christie Hospital, Manchester, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital, Nottingham, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - North Glasgow University Hospitals NHS Trust, Glasgow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simoes R, Gulliford S, Seddon B, Dehbi HM, Robinson M, Forsyth S, Hughes A, Gaunt P, Nguyen TG, Elston S, Mohammed K, Zaidi S, Miles E, Hoskin P, Harrington K, Miah A. Predicting radiotherapy response, Toxicities and quality-of-life related functional outcomes in soft tissue sarcoma of the extremities (PredicT) using dose-volume constraints development: a study protocol. BMJ Open. 2024 Aug 9;14(8):e083617. doi: 10.1136/bmjopen-2023-083617. PMID 39122389
- See also: Clinical trial summary from Cancer Research UK — http://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-looking-at-the-size-of-the-radiotherapy-treatment-area-for-people-with-soft-tissue-sarcoma